CLINICAL TRIAL: NCT02286479
Title: Comparison of Loop Drainage and Primary Incision and Drainage Techniques in Patients With Cutaneous Abscess in the Emergency Department
Brief Title: Comparison of Loop and Primary Incision&Drainage Techniques in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Ibrahim Ulas Ozturan, MD, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KOU KAEK 2014/259
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Skin Abscess
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incision and Drainage (Active Comparator): In the incision and drainage group, the abscesses are incised, irrigated by sterile solutions and drained conventionally.
  Interventions: Procedure: Incision and Drainage
- Loop drainage (Experimental): In the loop drainage group, two small incision are made on each side of abscess. The pus are drained and septations are seperated by a forceps. Abscess cavitary irrigated by sterile solution. Sterile, non-powder, non-latex surgical gloves cuff is inserted in one incision and taken out from the other insicion. Then two tips of cuff are tied loosely.
  Interventions: Procedure: Loop drainage

INTERVENTIONS:
Procedure: Incision and Drainage — In the incision and drainage group, the abscesses are incised, irrigated by sterile solutions and drained conventionally.
  Arms: Incision and Drainage
Procedure: Loop drainage — In the loop drainage group, two small incision are made on each side of abscess. The pus are drained and septations are seperated by a forceps. Abscess cavitary irrigated by sterile solution. Sterile, non-powder, non-latex surgical gloves cuff is inserted in one incision and taken out from the other insicion. Then two tips of cuff are tied loosely.
  Arms: Loop drainage

SUMMARY:
Skin abscesses are among the most common soft tissue infections cause emergency room visits frequently. Management of abscess drainage and prevent further complications are important entities for emergency physicians. Historically primary incision and drainage (I&D) technique has found very effective method of abscess drainage, however a novel technique loop drainage holds promising. The purpose of our study is comparison efficacy of I&D and loop drainage techniques in patients with cutaneous abscess.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting to Kocaeli University Emergency Department with cutaneous abscess.
* Providing written informed consent.

Exclusion Criteria:

* Under 18 years of age.
* Immunosuppressive patients.
* Using medications have effects on wound healing.
* Abscess is not recognizable by bedside ultrasound.
* Lidocaine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Abscess Resolution | 7 days

SECONDARY OUTCOMES:
Procedure Time | intraoperative

OTHER OUTCOMES:
Procedure Pain Intensity | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Medical Faculty Emergency Medicine Department, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ozturan IU, Dogan NO, Karakayali O, Ozbek AE, Yilmaz S, Pekdemir M, Suner S. Comparison of loop and primary incision & drainage techniques in adult patients with cutaneous abscess: A preliminary, randomized clinical trial. Am J Emerg Med. 2017 Jun;35(6):830-834. doi: 10.1016/j.ajem.2017.01.036. Epub 2017 Jan 22. PMID 28162873